CLINICAL TRIAL: NCT04502056
Title: Covid-19 Messaging to Underserved Communities - 2nd Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Massachusetts General Hospital (Other); Stanford University (Other); Yale University (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Esther Duflo, Abdul Latif Jameel Professor of Poverty Alleviation and Development Economics, MIT; Co-Director, Abdul Latif Jameel Poverty Action Lab, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2029880
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- AMA RI - B- B - R (Experimental): Respondents will be randomized to an AMA statement acknowledging racial injustice read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: Racial Inequality Highlighted
- AMA RI - B - B - N (Experimental): Respondents will be randomized to an AMA statement acknowledging racial injustice read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: No Racial Inequality Highlighting
- AMA RI - W - W - R (Experimental): Respondents will be randomized to an AMA statement acknowledging racial injustice read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: Racial Inequality Highlighted; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos
- AMA RI - W - W - N (Experimental): Respondents will be randomized to an AMA statement acknowledging racial injustice read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos; Behavioral: No Racial Inequality Highlighting
- AMA DP - B- B - R (Experimental): Respondents will be randomized to an AMA statement acknowledging drug pricing read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will include information on the disproportionate impact on communities of color .
  Interventions: Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: Racial Inequality Highlighted; Behavioral: AMA Acknowledgement Drug Pricing
- AMA DP - B- B - N (Experimental): Respondents will be randomized to an AMA statement acknowledging drug pricing read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: AMA Acknowledgement Drug Pricing; Behavioral: No Racial Inequality Highlighting
- AMA DP - W- W - R (Experimental): Respondents will be randomized to an AMA statement acknowledging drug pricing read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: Racial Inequality Highlighted; Behavioral: AMA Acknowledgement Drug Pricing; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos
- AMA DP - W- W - N (Experimental): Respondents will be randomized to an AMA statement acknowledging drug pricing read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Interventions: Behavioral: AMA Acknowledgement Drug Pricing; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos; Behavioral: No Racial Inequality Highlighting
- Control: AMA RI - B - B (Placebo Comparator): Respondents will be randomized to an AMA statement acknowledging racial injustice read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - No message on Covid-19 will be shown.
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: Placebo videos
- Control: AMA RI - W - W (Placebo Comparator): Respondents will be randomized to an AMA statement acknowledging racial injustice read by a white individual. The messenger / doctor in the follow-up AMA videos will also be white - No message on Covid-19 will be shown.
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  White Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a white sender in acknowledgment of AMA
  Interventions: Behavioral: Acknowledgement Racial Injustice AMA; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos; Behavioral: Placebo videos
- Control: AMA DP - B - B (Placebo Comparator): Respondents will be randomized to an AMA statement acknowledging drug pricing read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - No message on Covid-19 will be shown.
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  Interventions: Behavioral: African American Sender Acknowledgement; Behavioral: African American Sender in Informational Videos.; Behavioral: AMA Acknowledgement Drug Pricing; Behavioral: Placebo videos
- Control: AMA DP - W - W (Placebo Comparator): Respondents will be randomized to an AMA statement acknowledging drug pricing read by a white individual. The messenger / doctor in the follow-up AMA videos will also be white - No message on Covid-19 will be shown.
  White Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a white sender in acknowledgment of AMA
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  Interventions: Behavioral: AMA Acknowledgement Drug Pricing; Behavioral: White Sender in Acknowledgement; Behavioral: White Sender in Informational Videos; Behavioral: Placebo videos

INTERVENTIONS:
Behavioral: Acknowledgement Racial Injustice AMA — Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  Arms: AMA RI - B - B - N; AMA RI - B- B - R; AMA RI - W - W - N; AMA RI - W - W - R; Control: AMA RI - B - B; Control: AMA RI - W - W
Behavioral: African American Sender Acknowledgement — Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  Arms: AMA DP - B- B - N; AMA DP - B- B - R; AMA RI - B - B - N; AMA RI - B- B - R; Control: AMA DP - B - B; Control: AMA RI - B - B
Behavioral: African American Sender in Informational Videos. — Investigators will vary the sender of the informational covid-19 videos. In this arm, participants receive a African American sender in informational videos.
  Arms: AMA DP - B- B - N; AMA DP - B- B - R; AMA RI - B - B - N; AMA RI - B- B - R; Control: AMA DP - B - B; Control: AMA RI - B - B
Behavioral: Racial Inequality Highlighted — Investigators will include information on race-specific covid-19 cases and deaths in one variation in the messaging. In this arm, participants receive disproportionate race-specific Covid-19 facts
  Arms: AMA DP - B- B - R; AMA DP - W- W - R; AMA RI - B- B - R; AMA RI - W - W - R
Behavioral: AMA Acknowledgement Drug Pricing — Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  Arms: AMA DP - B- B - N; AMA DP - B- B - R; AMA DP - W- W - N; AMA DP - W- W - R; Control: AMA DP - B - B; Control: AMA DP - W - W
Behavioral: White Sender in Acknowledgement — Investigators will also vary the messenger of the acknowledgement sender. In this arm, participants receive a white sender in the acknowledgement
  Arms: AMA DP - W- W - N; AMA DP - W- W - R; AMA RI - W - W - N; AMA RI - W - W - R; Control: AMA DP - W - W; Control: AMA RI - W - W
Behavioral: White Sender in Informational Videos — Investigators will vary the messenger of the informational covid-19 videos. In this arm, participants receive white sender in the informational video
  Arms: AMA DP - W- W - N; AMA DP - W- W - R; AMA RI - W - W - N; AMA RI - W - W - R; Control: AMA DP - W - W; Control: AMA RI - W - W
Behavioral: No Racial Inequality Highlighting — In this arm, the disproportionate burden of Covid-19 on communities of color will not be highlighted
  Arms: AMA DP - B- B - N; AMA DP - W- W - N; AMA RI - B - B - N; AMA RI - W - W - N
Behavioral: Placebo videos — Videos not related to covid-19 will be shown
  Arms: Control: AMA DP - B - B; Control: AMA DP - W - W; Control: AMA RI - B - B; Control: AMA RI - W - W

SUMMARY:
The aim of the study is to build off results from our first experiment (NCT04371419) , and test whether messages that acknowledge racial injustice on behalf of institutions affect the retention of knowledge and movement of beliefs and behavior with respect to Covid-19. The investigators will also test the effect of concordance of providers and whether highlighting the unequal burden of the disease has additional effects on knowledge, beliefs and behavior regarding covid-19. The sample will include African American and white adult Americans and oversample those with less than a college degree.

DETAILED DESCRIPTION:
Recent data have shown that covid19 is disproportionately infecting and killing African Americans and Latinx people in the United States. Moreover, since our last experiment, the killing of George Floyd by Minnesota police has raised awareness of structural racism in the United States.

The aim of the study is to build off results from our first experiment (NCT04371419) , and test whether messages that acknowledge racial injustice on behalf of institutions affect the retention of knowledge and movement of beliefs and behavior with respect to Covid-19. The investigators will also test the effect of concordance of providers and whether highlighting the unequal burden of the disease has additional effects on knowledge, beliefs and behavior regarding covid-19.The sample will include African American and white adult Americans and oversample those with less than a college degree.

ELIGIBILITY:
Inclusion Criteria:

* adults who self-identify as African American or white.
* an oversample of individuals with less than a college education

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20460 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL North America, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Torres C, Ogbu-Nwobodo L, Alsan M, Stanford FC, Banerjee A, Breza E, Chandrasekhar AG, Eichmeyer S, Karnani M, Loisel T, Goldsmith-Pinkham P, Olken BA, Vautrey PL, Warner E, Duflo E; COVID-19 Working Group. Effect of Physician-Delivered COVID-19 Public Health Messages and Messages Acknowledging Racial Inequity on Black and White Adults' Knowledge, Beliefs, and Practices Related to COVID-19: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2117115. doi: 10.1001/jamanetworkopen.2021.17115. PMID 34259846

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: AMA RI - B- B - R: Respondents will be randomized to an AMA statement acknowledging racial injustice read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will include information on the disproportionate impact on communities of color .
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  African American Sender in Informational Videos.: Investigators will vary the sender of the informational covid-19 videos. In this arm, participants receive a African American sender in informational videos.
  Racial Inequality Highlighted: Investigators will include information on race-specific covid-19 cases and deaths in one variation in the messaging. In this arm, participants receive disproportionate race-specific Covid-19 facts
- Intervention: AMA RI - B - B - N: Respondents will be randomized to an AMA statement acknowledging racial injustice read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  African American Sender in Informational Videos.: Investigators will vary the sender of the informational covid-19 videos. In this arm, participants receive a African American sender in informational videos.
  No Racial Inequality Highlighting: In this arm, the disproportionate burden of Covid-19 on communities of color will not be highlighted
- Intervention: AMA RI - W - W - R: Respondents will be randomized to an AMA statement acknowledging racial injustice read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will include information on the disproportionate impact on communities of color.
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  Racial Inequality Highlighted: Investigators will include information on race-specific covid-19 cases and deaths in one variation in the messaging. In this arm, participants receive disproportionate race-specific Covid-19 facts
  White Sender in Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm, participants receive a white sender in the acknowledgement
  White Sender in Informational Videos: Investigators will vary the messenger of the informational covid-19 videos. In this arm, participants receive white sender in the informational video
- Intervention: AMA RI - W - W - N: Respondents will be randomized to an AMA statement acknowledging racial injustice read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  Acknowledgement Racial Injustice AMA: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants will receive a AMA statement on racial injustice.
  White Sender in Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm, participants receive a white sender in the acknowledgement
  White Sender in Informational Videos: Investigators will vary the messenger of the informational covid-19 videos. In this arm, participants receive white sender in the informational video
  No Racial Inequality Highlighting: In this arm, the disproportionate burden of Covid-19 on communities of color will not be highlighted
- Intervention: AMA DP - B- B - R: Respondents will be randomized to an AMA statement acknowledging drug pricing read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will include information on the disproportionate impact on communities of color .
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  African American Sender in Informational Videos.: Investigators will vary the sender of the informational covid-19 videos. In this arm, participants receive a African American sender in informational videos.
  Racial Inequality Highlighted: Investigators will include information on race-specific covid-19 cases and deaths in one variation in the messaging. In this arm, participants receive disproportionate race-specific Covid-19 facts
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
- Intervention: AMA DP - B- B - N: Respondents will be randomized to an AMA statement acknowledging drug pricing read by an African American individual. The messenger / doctor in the follow-up AMA videos will also be African American - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  African American Sender Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm participants receive a African American sender in acknowledgment of AMA
  African American Sender in Informational Videos.: Investigators will vary the sender of the informational covid-19 videos. In this arm, participants receive a African American sender in informational videos.
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  No Racial Inequality Highlighting: In this arm, the disproportionate burden of Covid-19 on communities of color will not be highlighted
- Intervention: AMA DP - W- W - R: Respondents will be randomized to an AMA statement acknowledging drug pricing read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will include information on the disproportionate impact on communities of color.
  Racial Inequality Highlighted: Investigators will include information on race-specific covid-19 cases and deaths in one variation in the messaging. In this arm, participants receive disproportionate race-specific Covid-19 facts
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  White Sender in Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm, participants receive a white sender in the acknowledgement
  White Sender in Informational Videos: Investigators will vary the messenger of the informational covid-19 videos. In this arm, participants receive white sender in the informational video
- Intervention: AMA DP - W- W - N: Respondents will be randomized to an AMA statement acknowledging drug pricing read by a white individual. The messenger / doctor in the follow-up AMA videos will be white - the message on Covid-19 will not include information on the disproportionate impact on communities of color.
  AMA Acknowledgement Drug Pricing: Investigators will examine whether acknowledgements of racial inequality are helpful towards improving knowledge retention and behaviors associated with the intervention among participants. In this arm, participants receive AMA information on drug pricing
  White Sender in Acknowledgement: Investigators will also vary the messenger of the acknowledgement sender. In this arm, participants receive a white sender in the acknowledgement
  White Sender in Informational Videos: Investigators will vary the messenger of the informational covid-19 videos. In this arm, participants receive white sender in the informational video
  No Racial Inequality Highlighting: In this arm, the disproportionate burden of Covid-19 on communities of color will not be highlighted
Period: Overall Study
Arm/Group | Intervention: AMA RI - B- B - R | Intervention: AMA RI - B - B - N | Intervention: AMA RI - W - W - R | Intervention: AMA RI - W - W - N | Intervention: AMA DP - B- B - R | Intervention: AMA DP - B- B - N | Intervention: AMA DP - W- W - R | Intervention: AMA DP - W- W - N | Control: AMA RI - B - B | Control: AMA RI - W - W | Control: AMA DP - B - B | Control: AMA DP - W - W
Started | 2046 | 2044 | 2045 | 2046 | 2044 | 2052 | 2046 | 2043 | 1026 | 1025 | 1023 | 1020
Completed the Knowledge Questions, Included for the Knowledge Gaps Analysis | 1859 | 1881 | 1879 | 1886 | 1846 | 1877 | 1888 | 1883 | 947 | 942 | 946 | 928
Completed the Entire Survey, Included for All Analysis Besides Knowledge Gaps, Except Follow-up | 1799 | 1828 | 1830 | 1835 | 1792 | 1820 | 1821 | 1844 | 914 | 912 | 928 | 900
Completed the Follow-up Survey | 608 | 607 | 591 | 601 | 631 | 598 | 607 | 607 | 301 | 313 | 291 | 316
Completed (Participants who completed follow-up and have no missing on baseline observables, included for follow-up analysis) | 604 | 602 | 586 | 597 | 626 | 596 | 605 | 603 | 298 | 311 | 288 | 614
Not Completed | 1442 | 1442 | 1459 | 1449 | 1418 | 1456 | 1441 | 1440 | 728 | 714 | 735 | 406

BASELINE CHARACTERISTICS:
Population: Any intervention was indeed an arm that included each sub arm of different types of message that we tested against a control and pre-specified in our study protocol and analysis plan to combine arms for analysis.
Groups:
- Intervention: Participants who are assigned to any intervention groups
- Control: Participants who are assigned to a control group
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 14145 | 3544 | 17689
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.20 (17.83) | 40.30 (17.73) | 40.22 (17.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7907 | 1973 | 9880
  Male | 6238 | 1571 | 7809
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6303 | 1576 | 7879
  White | 7842 | 1968 | 9810
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast, United States | 2424 | 600 | 3024
  United States: Midwest, United States | 3114 | 770 | 3884
  United States: South, United States | 6397 | 1649 | 8046
  United States: West, United States | 2210 | 525 | 2735
High school graduate [Count of Participants; unit: Participants] | 12009 | 3007 | 15016
Household income above 60k [Count of Participants; unit: Participants] | 3356 | 850 | 4206
Party Affiliation [Count of Participants; unit: Participants]
  Democrat | 5594 | 1383 | 6977
  Republican | 3494 | 882 | 4376
  Independent | 5057 | 1279 | 6336
Preventive practices: mask in (always) [Count of Participants; unit: Participants] | 9648 | 2458 | 12106
Preventive practices: mask out (always) [Count of Participants; unit: Participants] | 4408 | 1109 | 5517
Preventive practices: wash hands (always) [Count of Participants; unit: Participants] | 8688 | 2091 | 10779
Preventive practices: distance (always) [Count of Participants; unit: Participants] | 7571 | 1890 | 9461

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate for Knowledge Gaps: Control vs. Any Intervention
Description: Participants were asked to identify ways to prevent COVID-19 spread and identify four common symptoms. The incidence rate for knowledge gaps is the count of knowledge gaps divided by the maximum possible count: 10.
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of knowledge gaps
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14999 | 3763
proportion of knowledge gaps | 0.214 [0.211 to 0.217] | 0.241 [0.235 to 0.246]

2. Primary Outcome: Incidence Rate for Knowledge Gaps: Control vs. Any Intervention - Follow up
Description: Participants were asked to identify ways to prevent COVID-19 spread and identify four common symptoms. Incidence rate for knowledge gaps is the count of knowledge gaps divided by the maximum possible count: 10.
Time Frame: The outcome was measured at a follow-up within 2 weeks following the intervention
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of knowledge gaps
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4819 | 1211
proportion of knowledge gaps | 0.241 [0.238 to 0.244] | 0.250 [0.243 to 0.256]

3. Primary Outcome: Incidence Rate for Information-seeking Behavior: Control vs. Any Intervention
Description: Participants were offered the option of requesting additional information on COVID-19 related resources by clicking on up to five links that included more content. We measured "information seeking behavior" as the number of links for which participants expressed interest, a count variable between 0 (lowest information seeking behavior) and 5 (greatest information seeking behavior). Incidence rate for interest in links is the count of links demanded divided by the maximum possible count: 5.
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of links
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14569 | 3654
proportion of links | 0.338 [0.332 to 0.344] | 0.320 [0.308 to 0.332]

4. Primary Outcome: Incidence Rate - Safety Gap Score: Control vs. Any Intervention
Description: Participants were asked about how often they engaged in four behaviors of interest: if they wore a mask indoors/outdoors; if they washed their hands; if they followed social distancing guidelines. The safety gap index takes values of 0 (if a participant reported that they always practiced the four behaviors of interest) up to 4 (none). Incidence rate for safety gaps is the count of safety gaps divided by the maximum possible count: 4.
Time Frame: The outcome was measured at a follow-up within 2 weeks following the intervention.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of safety gaps
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4823 | 1212
proportion of safety gaps | 0.450 [0.440 to 0.460] | 0.465 [0.445 to 0.484]

5. Primary Outcome: Willingness to Pay (WTP) for Masks: Control vs. Any Intervention
Description: WTP: the participants will be asked to choose between two masks vs an unrestricted gift card. They will be asked what amount of gift card would make them just as happy to receive two mask versus the gift card.
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollar
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13399 | 3360
dollar | 14.580 [14.148 to 14.741] | 14.072 [13.762 to 14.382]

6. Primary Outcome: Incidence Rate Ratio (IRR) - Knowledge Gap
Description: Participants were asked to identify ways to prevent COVID-19 spread and identify four common symptoms. The incidence rate for knowledge gaps is the count of knowledge gaps divided by the maximum possible count: 10. The incidence rate ratio compares the incidence rate of participants in Arm A vs. Arm B within the intervention group (i.e. those who received covid-19-related videos), within in the control group (i.e. those who saw placebo videos), or across the intervention and control group. Arms A and B are described in each Arm/Group Title. The overall number of participants analyzed is all equal across 6 arms/groups because the outcome measure data presented below came from a single negative binomial regression.
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: Arms were combined to assess the differential effectiveness of each unique video message by comparing participants in Arm A vs. Arm B, since Arm A cut across several other studies:
  1. within the intervention group; or
  2. within the control group; or
  3. across the intervention and control groups.
  Arms A and B are described in each Arm/Group Title.
Measure: Number (95% Confidence Interval); unit: ratio
Groups:
- Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B): The relative IRR for intervention participants who saw a message delivered by a Black doctor and saw covid-19-related messages vs. those who did not see either or neither of the messages.
- Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B): The relative IRR for intervention participants who saw the AMA anti-racism treatment and saw covid-19-related messages vs. those who did not see either or neither of the messages.
- Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B): The relative IRR for intervention participants who saw the message on the relative incidence of COVID-19 among Black and white individuals and saw covid-19-related messages vs. those who did not see either or neither of the messages.
- Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B): The relative IRR for intervention participants who saw a Black doctor vs. white doctor
- Within Control Group: AMA Anti-racism vs. Either/Neither: The relative IRR for intervention participants who saw the AMA anti-racism treatment vs. those who saw the placebo message.
- Intervention Group vs. Control Group: The relative IRR for intervention participants who saw covid-related messages vs. those who did not see any covid-19 related messages.
Arm/Group | Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B) | Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B) | Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Control Group: AMA Anti-racism vs. Either/Neither | Intervention Group vs. Control Group
Number analyzed (Participants) | 18762 | 18762 | 18762 | 18762 | 18762 | 18762
ratio | 1.01 [0.96 to 1.06] | 0.99 [0.94 to 1.04] | 1.01 [0.98 to 1.03] | 0.99 [0.95 to 1.04] | 0.99 [0.95 to 1.03] | 0.89 [0.85 to 0.93]

7. Primary Outcome: Incidence Rate Ratio (IRR) - Knowledge Gap - Follow up
Description: as for outcome 6
Time Frame: The outcome was measured at a follow-up within 2 weeks following the intervention
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B) | Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B) | Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Control Group: AMA Anti-racism vs. Either/Neither | Intervention Group vs. Control Group
Number analyzed (Participants) | 6030 | 6030 | 6030 | 6030 | 6030 | 6030
ratio | 0.98 [0.90 to 1.07] | 0.98 [0.90 to 1.07] | 1.01 [0.98 to 1.05] | 1.01 [0.94 to 1.09] | 0.98 [0.91 to 1.06] | 0.97 [0.90 to 1.04]

8. Primary Outcome: Incidence Rate Ratio (IRR) - Information-seeking Behavior
Description: Participants were offered the option of requesting additional information on COVID-19 related resources by clicking on up to 5 links that included more content. We measured "information seeking behavior" as the number of links for which participants expressed interest, a count variable between 0 (lowest information seeking behavior) and 5 (greatest information seeking behavior). Incidence rate for interest in links is the count of links demanded divided by the maximum possible count: 5. The incidence rate ratio compares the incidence rate of participants in Arm A vs. Arm B within the intervention group (i.e. those who received covid-19-related videos), within in the control group (i.e. those who saw placebo videos), or across the intervention and control group. Arms A and B are described in each Arm/Group Title. The overall number of participants analyzed is all equal across 6 arms/groups because the outcome measure data presented below came from a single negative binomial regression.
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B) | Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B) | Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Control Group: AMA Anti-racism vs. Either/Neither | Intervention Group vs. Control Group
Number analyzed (Participants) | 18223 | 18223 | 18223 | 18223 | 18223 | 18223
ratio | 1.04 [0.95 to 1.14] | 1.03 [0.93 to 1.13] | 1.02 [0.98 to 1.07] | 0.96 [0.89 to 1.05] | 0.97 [0.89 to 1.05] | 1.01 [0.93 to 1.10]

9. Primary Outcome: Incidence Rate Ratio (IRR) - Safety Gap Score
Description: Participants were asked about how often they engaged in four behaviors of interest: if they wore a mask indoors/outdoors; if they washed their hands; if they followed social distancing guidelines. The safety gap index takes values of 0 (if a participant reported that they always practiced the four behaviors of interest) up to 4 (none). Incidence rate for safety gaps is the count of safety gaps divided by the maximum possible count: 4. The incidence rate ratio compares the incidence rate of participants in Arm A vs. Arm B within the intervention group (i.e. those who received covid-19-related videos), within in the control group (i.e. those who saw placebo videos), or across the intervention and control group. Arms A and B are described in each Arm/Group Title. The overall number of participants analyzed is all equal across 6 arms/groups because the outcome measure data presented below came from a single negative binomial regression.
Time Frame: The outcome was measured at a follow-up within 2 weeks following the intervention.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B) | Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B) | Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Control Group: AMA Anti-racism vs. Either/Neither | Intervention Group vs. Control Group
Number analyzed (Participants) | 6035 | 6035 | 6035 | 6035 | 6035 | 6035
ratio | 1.04 [0.95 to 1.14] | 1.03 [0.93 to 1.12] | 1.01 [0.97 to 1.05] | 0.97 [0.89 to 1.05] | 0.95 [0.87 to 1.03] | 0.93 [0.86 to 1.01]

10. Primary Outcome: OLS Regression Coefficients - Willingness to Pay (WTP) for Masks
Description: WTP: the participants will be asked to choose between two masks vs an unrestricted gift card. They will be asked what amount of gift card would make them just as happy to receive two mask versus the gift card. The regression coefficients compares the incidence rate of participants in Arm A vs. Arm B within the intervention group (i.e. those who received covid-19-related videos), within in the control group (i.e. those who saw placebo videos), or across the intervention and control group. Arms A and B are described in each Arm/Group Title. The overall number of participants analyzed is all equal across 6 arms/groups because the outcome measure data presented below came from a single ordinary least squares (OLS) regression for WTP masks).
Time Frame: The outcome was measured immediately following the intervention in the baseline survey.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: dollar
Arm/Group | Within Intervention Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Intervention Group: AMA Anti-racism (Arm A) vs. Either/Neither (Arm B) | Within Intervention Group: Doctor Racial Disparity (Arm A) vs. Either/Neither (Arm B) | Within Control Group: Black Physician (Arm A) vs. White Physician (Arm B) | Within Control Group: AMA Anti-racism vs. Either/Neither | Intervention Group vs. Control Group
Number analyzed (Participants) | 16759 | 16759 | 16759 | 16759 | 16759 | 16759
dollar | -0.21 [-0.91 to 0.49] | -0.29 [-0.99 to 0.41] | 0.07 [-0.24 to 0.39] | 0.17 [-0.45 to 0.80] | 0.32 [-0.30 to 0.95] | 0.71 [0.09 to 1.34]

ADVERSE EVENTS:
Time Frame: 31 days
Arm/Group | Intervention: AMA RI - B- B - R | Intervention: AMA RI - B - B - N | Intervention: AMA RI - W - W - R | Intervention: AMA RI - W - W - N | Intervention: AMA DP - B- B - R | Intervention: AMA DP - B- B - N | Intervention: AMA DP - W- W - R | Intervention: AMA DP - W- W - N | Control: AMA RI - B - B | Control: AMA RI - W - W | Control: AMA DP - B - B | Control: AMA DP - W - W
All-Cause Mortality (participants affected / at risk) | 0/2046 | 0/2044 | 0/2045 | 0/2046 | 0/2044 | 0/2052 | 0/2046 | 0/2043 | 0/1026 | 0/1025 | 0/1023 | 0/1020
Serious Adverse Events (participants affected / at risk) | 0/2046 | 0/2044 | 0/2045 | 0/2046 | 0/2044 | 0/2052 | 0/2046 | 0/2043 | 0/1026 | 0/1025 | 0/1023 | 0/1020
Other Adverse Events (participants affected / at risk) | 0/2046 | 0/2044 | 0/2045 | 0/2046 | 0/2044 | 0/2052 | 0/2046 | 0/2043 | 0/1026 | 0/1025 | 0/1023 | 0/1020

LIMITATIONS AND CAVEATS:
1. It was conducted online, and the participants may not be representative of the population with less than a college degree, since they have access to the internet and are used to participating in online studies; 2. Participants' preventive health behaviors were not directly observed; 3. Outcomes might be subject to social desirability bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT04502056/Prot_SAP_000.pdf